CLINICAL TRIAL: NCT02689739
Title: Lower-extremity Blood fl ow and Velocity in Obese vs Nonobese Pregnant Women
Brief Title: Validation of Ultrasound in Predicting a Low Lying Placenta Throughout Pregnancy
Status: Withdrawn | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0143
Record Dates: First submitted 2016-02-13; First posted 2016-02-24 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2019-03

CONDITIONS: Pregnancy; Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese Pregnant cohort: Women will be consented to participate and then separated into a study group of obese women (BMI >/= 30).
  Interventions: Procedure: venous duplex ultrasound
- Non-obese Pregnant cohort: This will be the control group of non-obese women (BMI <30).
  Interventions: Procedure: venous duplex ultrasound

INTERVENTIONS:
Procedure: venous duplex ultrasound — Venous duplex ultrasound

SUMMARY:
This is a prospective observational study comparing venous Doppler flow in the lower extremities of pregnant women. Pregnant women with a BMI >/= 30 will be compared to those with a BMI < 30.

DETAILED DESCRIPTION:
Study Outcome Measurement and Ascertainment:

Data will be collected from data in EPIC and UTMB electronic medical records. This information will include:

1. Maternal demographic data, medical, family, personal, social and surgical history
2. Maternal pre-pregnancy weight and height
3. Maternal weight at time of delivery
4. Maternal weight on post-operative day 1
5. Gestational age at delivery, infant gender, birth weight, placental weight, delivery method, and complications through 6 weeks postpartum.

Venous hemodynamics will be obtained using venous duplex ultrasound. 1. Peak, mean, and minimum flow velocities and diameter will be obtained. Calculations of venous velocity amplitude, cross-sectional area, and shear stress will be made from the data collected.

Study Procedures:

This is a prospective study using duplex ultrasound techniques to characterize venous flow in obese and non-obese pregnant patients. Women will be consented to participate and then separated into a study group of obese women (BMI >/= 30) and a control group of non-obese women (BMI <30). These women will be admitted to Labor and Delivery for management of pregnancy. The Doppler US will then be performed by trained staff on the lower extremity. The flow data described above will be measured and compared between the two groups. Additional measurements will be collected during hospitalization.

Criteria for Inclusion of Subjects:

-Age >/= 18 years of age, planned delivery at John Sealy Hospital (JSH)

Criteria for Exclusion of Subjects:

* <18 years of age
* Personal history of VTE, regardless of etiology
* Development of VTE during this pregnancy -History of thrombophilia, bleeding disorder marked varicosities, history of recurrent stillbirth, intrauterine growth restriction
* Any indication for emergency delivery
* Known major fetal abnormality or genetic syndrome

Sources of Research Material:

The sources of data to be used include maternal medical records from EPIC as well as the data obtained from the venous ultrasound.

Recruitment Methods and Consenting Process:

The subjects will be pregnant women who plan a delivery at JSH. Subjects will be consented by study personnel. Patients will not receive any monetary gain. They will understand that this is voluntary and will not affect their care.

Potential Risks:

The Doppler velocimetry is the modality that has been used in pregnancy to assess for the presence of DVT, thus, the safety has been assessed and widely studied. This poses minimum risk to the mother or to the fetus.

Subject Safety and Data Monitoring:

This study does not place subjects at risk of their safety. This modality is well studied to be safe in pregnancy.

Data monitoring will be performed only by study personnel. Data may be assessed prior to the study being completed to assess to see if statistical analysis reveals any difference and if the study can be stopped early.

Procedures to Maintain Confidentiality:

Data will only be viewed by study personnel. The data will then be de-identified and a study number will be assigned to each patient. The patient's identity will then be secured on an UTMB encrypted laptop device and a hard copy stored in the locked file cabinet in the locked office of the investigator.

Potential Benefits:

There are no benefits to subjects participating in the study. By gathering the information of duplex velocimetry in both the obese and non-obese population we can determine if there is a change in the velocimetry in this at risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years of age, planned delivery at John Sealy Hospital (JSH)

Exclusion Criteria:

* <18 years of age
* Personal history of VTE, regardless of etiology
* Development of VTE during this pregnancy -History of thrombophilia, bleeding disorder marked varicosities, history of recurrent stillbirth, intrauterine growth restriction
* Any indication for emergency delivery
* Known major fetal abnormality or genetic syndrome

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a prospective study comparing venous Doppler flow in the lower extremities of pregnant women. Pregnant women with a BMI >/= 30 will be compared to those with a BMI < 30 who deliver at UTMB.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change in venous duplex velocity | On admission for delivery of the infant and postpartum day 1 and 2
  To assess if the increased risk of venous thromboembolism is observed in obese versus non-obese pregnant patients is due to compromised flow in the lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Olson, MD, Study Director — UTMB
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share data.